CLINICAL TRIAL: NCT04712396
Title: An Open-label, Fixed Sequence Study in Healthy Subjects to Assess the Pharmacokinetics of Capivasertib When Administered Alone and In Combination With Itraconazole
Brief Title: A Study to Assess How Itraconazole Affects the Uptake and Elimination of Capivasertib in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D3614C00004
Record Dates: First submitted 2020-12-15; First posted 2021-01-15 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Healthy Volunteers (Intended Indication: Metastatic Patients With Triple Negative or HR+ Breast Cancer, or Hormone Sensitive Prostate Cancer)
Keywords: Drug-Drug Interaction; Protein kinase inhibitor; Capivasertib; Itraconazole
MeSH Terms: interventions — capivasertib; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Capivasertib + Itraconazole (Experimental): Subjects will receive a single oral dose of capivasertib on Day 1 during treatment period 1, itraconazole on Days 3, 4, and 5 during treatment period 2, and single oral dose of capivasertib plus a dose of itraconazole on Day 6, followed by itraconazole alone on Day 7 during treatment period 3.
  Interventions: Drug: Capivasertib; Drug: Itraconazole

INTERVENTIONS:
Drug: Capivasertib — Subects will be administered single doses of capiversatib on Day 1 and Day 6.
Drug: Itraconazole — Subjects will be administered itraconazole twice daily on Day 3, followed by once daily doses in the morning for 4 days.

SUMMARY:
This study will be an open-label, fixed sequence study in healthy subjects (vasectomized males and females of non-childbearing potential), performed at a single study centre.

DETAILED DESCRIPTION:
The study will comprise:

* A screening period of maximum 21 days;
* A fixed sequence of 3 treatment periods: Treatment Period 1: Capivasertib only, Treatment Period 2: Itraconazole pre-treatment (run-in) period, and Treatment Period 3: Capivasertib and itraconazole in combination.
* A Follow-up Visit at 7 to 14 days after the last capivasertib PK sample in Treatment Period 3.

There will be no washout between Treatment Period 2 and Treatment Period 3. Each subject will be involved in the study for up to 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and female subjects aged 18 to 58 years with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative pregnancy test at screening and on admission to the study centre, must not be lactating and must be of non-childbearing potential, confirmed at screening.
* Male subjects must be vasectomized (at least 6 months prior to the Screening Visit), with documented post-procedural medical assessment of surgical success.
* Have a body mass index between 18 and 28 kg/m^2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
* Non-smoker, defined as a subject who has not smoked previously or who has discontinued smoking or the use of other nicotine/nicotine-containing products.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs; abnormalities in haematology, clinical chemistry, or urinalysis results, at screening or on admission to the study centre, as judged by the Investigator.
* Any clinically significant abnormalities in glucose metabolism, blood lipid profiles , liver enzymes , vital signs , and 12-lead electrocardiogram.
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg) or antibody to hepatitis B core antigen (anti-HBc), hepatitis C antibody (anti-HCV), and human immunodeficiency virus (HIV) antibody.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator.
* Positive screen for drugs of abuse, alcohol and/or cotinine at screening or on admission to the study centre.
* Subjects who have previously received capivasertib.
* Subject has a positive test result for Severe acute respiratory syndrome (SARS)-Coronavirus (CoV)-2 Reverse Transcriptase (RT)-Polymerase Chain Reaction (PCR) before randomization.
* Subject has clinical signs and symptoms consistent with corona virus disease 2019 (COVID-19) (e.g., fever, dry cough, dyspnoea, sore throat, anosmia/hyposmia, loss or reduced taste, and fatigue) or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.
* Subjects who are regularly exposed to the risk of COVID-19 infection as part of their daily life (e.g., health care professionals working in COVID-19 wards or at emergency departments).

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from zero to infinity (AUCinf) of capivasertib | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours after capivasertib dose on Day 1 and Day 6
  Assessment of AUCinf of capivasertib.
Maximum observed plasma (peak) drug concentration (Cmax) of capivasertib | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours after capivasertib dose on Day 1 and Day 6
  Assessment of Cmax of capivasertib.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUClast) of capivasertib and its major metabolite (AZ14102143) | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours after capivasertib dose on Day 1 and Day 6
  Assessment of AUClast of capivasertib and its major metabolite (AZ14102143).
Time delay between drug administration and the first observed concentration in plasma (tlag) of capivasertib | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours after capivasertib dose on Day 1 and Day 6
  Assessment of tlag of capivasertib.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) of capivasertib and its major metabolite (AZ14102143) | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours after capivasertib dose on Day 1 and Day 6
  Assessment of tmax of capivasertib and its major metabolite (AZ14102143).
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration time curve (t½λz) of capivasertib and its major metabolite (AZ14102143) | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours after capivasertib dose on Day 1 and Day 6
  Assessment of t½λz of capivasertib and its major metabolite (AZ14102143).
Terminal elimination rate constant (λz) of capivasertib and its major metabolite (AZ14102143) | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours after capivasertib dose on Day 1 and Day 6
  Assessment of λz of capivasertib and its major metabolite (AZ14102143).
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) of capivasertib | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours after capivasertib dose on Day 1 and Day 6
  Assessment of CL/F of capivasertib.
Volume of distribution (apparent) at steady state following extravascular administration (Vz/F) (based on terminal phase) of capivasertib | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours after capivasertib dose on Day 1 and Day 6
  Assessment of Vz/F of capivasertib.
AUCinf of major metabolite (AZ14102143) of capivasertib | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours after capivasertib dose on Day 1 and Day 6
  Assessment of AUCinf of major metabolite (AZ14102143) of capivasertib.
Cmax of major metabolite (AZ14102143) of capivasertib | Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours after capivasertib dose on Day 1 and Day 6
  Assessment of Cmax of major metabolite (AZ14102143) of capivasertib.
Number of subjects with serious and non-serious adverse events | From Screening until Follow-upVisit / Early Termination (7-14 days after last PK sample)
  Assessment of safety and tolerability of capivasertib alone and in combination with itraconazole.

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, Dr., Principal Investigator — Parexel
Locations (1):
- Research Site, Berlin, Germany